CLINICAL TRIAL: NCT06852690
Title: The Effect of Virtual Exercises on Glycemic Control, Body Composition, Psychological Status and Quality of Life in Type 2 Diabetic Patients
Brief Title: The Effect of Virtual Exercises on Glycemic Control and Body Composition in Type 2 Diabetic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Sabahattin Zaim University (Other)
Responsible Party: Principal Investigator, Kibar BZK, Investigator, Istanbul Sabahattin Zaim University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2023-07
Record Dates: First submitted 2025-02-06; First posted 2025-02-28 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Diabetes Mellitus Type 2
Keywords: diabetes, glycemic control, virtual reality, quality of life
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant
Masking Description: Virtual reality glasses and control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual reality glasses (Experimental): Patients with type 2 diabetes were planned to exercise for 10 minutes warm-up and 10 minutes cool down and 30 minutes exercise for 50 minutes in total
  Interventions: Other: exercise with virtual reality goggles
- Control group (No Intervention): Routine maintenance will be applied

INTERVENTIONS:
Other: exercise with virtual reality goggles — Exercise and smartwatch tracking for type 2 diabetics with virtual reality glasses
  Arms: Virtual reality glasses

SUMMARY:
This study was conducted to evaluate the effect of exercises with VR goggles in patients with type 2 diabetes.

The effect of exercise in virtual reality goggles on glycemic control, body composition, quality of life and psychological status.

DETAILED DESCRIPTION:
For virtual reality applications, a screen will be worn on the user's head that provides a three-dimensional visual image, thus creating a sense of space and depth. Blood glucose levels, vital signs and oxygen consumption capacity measurements will be monitored with the smart watch throughout the VR exercise application.

ELIGIBILITY:
Inclusion Criteria:

Being over 18 years old able to communicate Volunteering to participate in the research

Exclusion Criteria:

Those with psychiatric problems Being unconscious

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2023-07-28 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Glycemic Control Analysis | 3 months
  HbA1c levels of patients in the intervention and control groups will be checked
Analysis of Body Composition Values | 3 months
  Body analysis will be performed with a validated device. The patient will be measured before and after exercise and fat mass, lean mass, muscle mass, visceral fat ratio and basal metabolic rate will be measured by the device.
fat mass | 3 months
  patients will be tested for fat mass on the device
lean mass | 3 months
  patients will have a device to check their lean mass.
muscle mass | 3 months
  patients' muscle mass will be checked with the device
visceral fat content | 3 months
  patients will be tested for visceral fat with the device
basal metabolic rate | 3 months
  patients' basal metabolic rate will be monitored with the device

SECONDARY OUTCOMES:
Depression Anxiety Stress Scale | 3 months
  As the score of the answers to the questions increases, the level of depression, anxiety and stress increases. A score of 5 points or more in the depression sub-dimension, 4 points or more in anxiety, and 8 points or more in stress indicates that the individual has a related problem.
SF-36 Quality of Life Scale | 3 months
  The scale, which includes thirty-six statements, is a multi-item scale assessing 8 health concepts (physical function, physical role, fitness/fatigue, pain, general health perception, social function, emotional role, mental health) and 2 main topics (physical dimension and mental dimension).
Satisfaction Survey | 3 months
  There are 11 questions to evaluate the satisfaction of the patients about VR application and to question the conditions such as headache, dizziness, eye fatigue, disorientation, vertigo, loss of skin color, nausea and vomiting that may develop due to the use of virtual reality goggles.

CONTACTS AND LOCATIONS:
Locations (1):
- İstanbul Sabahattin Zaim Üniversitesi, Sağlık Bilimleri Fakültesi, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No